CLINICAL TRIAL: NCT04346303
Title: Intervention Feasibility and Outcomes Evaluation of Applying Short-term Interactive Video Games on Community Patients With Mental Disorders
Brief Title: Applying Short-term Interactive Video Games on Community Patients With Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202001106RIND
Record Dates: First submitted 2020-03-31; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-03

CONDITIONS: Psychiatry; Nursing
Keywords: Short-term Interactive Video Games; Community Patients with Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-term Interactive Video Games (Other): Short-term video games will be applied to patients with mental illness who are staying in communities. Games will be applied in a group-activity format with 8 to 12 patients in each session. The interventions will be conducted at a two sessions per week for a 3-week long period. There are 3 time points for data collection, including 2-weeks before the intervention, the week before the intervention, and the week after the intervention. Each patient will be his/her own controlled comparison.
  Interventions: Other: Short-term Interactive Video Games

INTERVENTIONS:
Other: Short-term Interactive Video Games — 1. Collect basic information through a structured questionnaire, which includes basic information, disease status, life style and other related information.
  2. Three data collections were performed, namely the baseline period (T0) and the pre-program (T1) two weeks later. Three weeks of intervention activities were provided twice a week, followed by a post-test ( post-program, T2).
  3. After a total of six times mentioned above, each 60 minutes of interactive video game intervention, the patient completed the activity feedback form, reflecting the feelings and feedback of participating in the activity.

SUMMARY:
The purpose of this study is to design prospective experiments before and after the test. The purpose is to explore whether short-term interactive video games can improve the motivation, interpersonal interaction, and physical and mental health of patients with mental illness in community rehabilitation homes. Samples of mentally ill patients from community rehabilitation homes (full-day rehabilitation institutions) in the northern region were collected using a structured questionnaire for the recipients, as follows:

1. Collect basic information through a structured questionnaire, which includes basic information, disease status, life style and other related information.
2. Three data collections were performed, namely the baseline period (T0) and the pre-program (T1) two weeks later. Three weeks of intervention activities were provided twice a week, followed by a post-test ( post-program, T2).
3. After a total of six times mentioned above, each 60 minutes of interactive video game intervention, the patient completed the activity feedback form, reflecting the feelings and feedback of participating in the activity.

DETAILED DESCRIPTION:
The purpose of this study is to design prospective experiments before and after the test. The purpose is to explore whether short-term interactive video games can improve the motivation, interpersonal interaction, and physical and mental health of patients with mental illness in community rehabilitation homes. Samples of mentally ill patients from community rehabilitation homes (full-day rehabilitation institutions) in the northern region were collected using a structured questionnaire for the recipients, as follows:

1. Collect basic information through a structured questionnaire, which includes basic information, disease status, life style and other related information.
2. Three data collections were performed, namely the baseline period (T0) and the pre-program (T1) two weeks later. Three weeks of intervention activities were provided twice a week, followed by a post-test ( post-program, T2).
3. After a total of six times mentioned above, each 60 minutes of interactive video game intervention, the patient completed the activity feedback form, reflecting the feelings and feedback of participating in the activity.

Primary Outcome Measure:

The changes of quality of life (WHOQOL-BREF: WHO Quality of Life: Brief form) After Short-term Interactive Video Games the changes of quality of life. This is a 28-items quality of life measurement to assess patient's quality of life.

[Time Frame: 5 Weeks]

Secondary Outcome Measures:

Body Mass Index Measuring height and weight [Time Frame: 5 Weeks]

Waist-hip ratio Measuring the ratio of waist to hip [Time Frame: 5 Weeks]

10-m walking time at comfortable Measuring the 10-m walking time at comfortable [Time Frame: 5 Weeks]

10-m walking time at maximum Measuring the 10-m walking time at maximum [Time Frame: 5 Weeks]

Get Up and Go test Measuring the Get Up and Go test [Time Frame: 5 Weeks]

5 times sit-to-stand test Measuring the 5 times sit-to-stand test [Time Frame: 5 Weeks]

Hierarchy of the Care Required This is a 18-item questionnaire to assess the patient's ADL and IADL as well as daily function.

[Time Frame: 5 Weeks]

CHQ-12 (Chinese Health Questionnaire) This is a 12-item scale to assess the patient's life stress indicating anxiety and depression symptoms.

[Time Frame: 5 Weeks]

Short FES-I (Chinese version of the Falls Efficacy Scale ) This is a 7-item scale to assess patient's vulnerability to fall. [Time Frame: 5 Weeks]

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis conforms to the international classification standards for the diagnosis of dysphoria or bipolar disorder.
* Be older than 20 years old.
* those who have a clear sense and can communicate.
* You can read the instructions carefully, and after you explain, you are willing to participate in the research plan and fill out the consent form.
* The judges of the researchers can independently answer the interview questionnaires of this research and perform short-term interactive video game players.
* At present, you can go out, make friends, take care of yourself, and fully exercise your rights. You have the full capacity of an adult and have not been restricted by any laws. Therefore, you do not need to obtain an additional legal agent to participate in this study Sign the consent form.

Exclusion Criteria:

* People with difficulties in cognitive understanding, such as those who cannot communicate or suffer from cognitive impairments, such as Alzheimer's disease.
* Those who have obvious obstacles to the physical function of their limbs, who are unable to participate in sports video games.
* Slow development or lack of moderate intelligence may affect the understanding of interviews or participation in activities.
* The physical and mental condition has been unstable in the past two weeks, such as instability of vital signs or obvious impaired sense of reality, obvious symptoms of delusions or hallucinations, etc., cannot be interviewed or coordinated with activities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of quality of life (WHOQOL-BREF: WHO Quality of Life: Brief form) | 5 Weeks
  After Short-term Interactive Video Games the changes of quality of life. This is a 28-items quality of life measurement to assess patient's quality of life.

SECONDARY OUTCOMES:
Body Mass Index | 5 Weeks
  Measuring height and weight
Waist-hip ratio | 5 Weeks
  Measuring the ratio of waist to hip
10-m walking time at comfortable | 5 Weeks
  Measuring the 10-m walking time at comfortable
10-m walking time at maximum | 5 Weeks
  Measuring the 10-m walking time at maximum
Get Up and Go test | 5 Weeks
  Measuring the Get Up and Go test
5 times sit-to-stand test | 5 Weeks
  Measuring the 5 times sit-to-stand test
Hierarchy of the Care Required | 5 Weeks
  This is a 18-item questionnaire to assess the patient's ADL and IADL as well as daily function.
CHQ-12 (Chinese Health Questionnaire) | 5 Weeks
  This is a 12-item scale to assess the patient's life stress indicating anxiety and depression symptoms.
Short FES-I (Chinese version of the Falls Efficacy Scale ) | 5 Weeks
  This is a 7-item scale to assess patient's vulnerability to fall.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Jung-Chen, PhD, Principal Investigator — National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No